CLINICAL TRIAL: NCT03482089
Title: Cystoprostatectomy Versus Radiotherapy Combined With Androgen Deprivation Therapy for the Treatment of Clinical T4 Prostate Cancer With Bladder Invasion: a Multicentre, Prospective, Open, Randomized Clinical Trial
Brief Title: Cystoprostatectomy Versus Radiotherapy Combined With ADT for the Treatment of cT4 Prostate Cancer With Bladder Invasion
Acronym: CRADT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Xiangya Hospital of Central South University (Other); Hubei Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZQ5208
Record Dates: First submitted 2018-03-18; First posted 2018-03-29 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystoprostatectomy (Experimental): (Open, laparoscopic or robot-assisted ) cystoprostatectomy with urinary diversion surgery and extended pelvic lymph node dissection; without adjuvant androgen deprivation therapy;
  Interventions: Procedure: Cystoprostatectomy
- Radiotherapy (Active Comparator): Radiotherapy by external beam radiotherapy (81 Gy，2.4-4 Gy per fraction over 4-6 weeks); with adjuvant androgen deprivation therapy for the least 3 years
  Interventions: Radiation: external beam radiotherapy

INTERVENTIONS:
Procedure: Cystoprostatectomy — Patients with bladder infiltrating T4 prostate cancer receive cystoprostatectomy with urinary diversion surgery and extended pelvic lymph node dissection
  Arms: Cystoprostatectomy
Radiation: external beam radiotherapy — Patients with bladder infiltrating T4 prostate cancer are treated with adjuvant androgen deprivation therapy
  Arms: Radiotherapy

SUMMARY:
Prostate cancer is the most common male cancer in global, which accounts for 19% of the total and poses great hazards to male health. Unfavorable factors including prostatic specific antigen (PSA) >20 ng/ml, Gleason score >8, and T3/4 are significantly associated with biological recurrence, metastatic progression and poor survival in prostate cancer. In clinical T4(cT4) prostate cancer with bladder invasion patients, symptoms of hematuria, urinary urgency, bladder outlet and ureteral obstruction, and pelvic pain led to a poor quality of life.

Radical prostatectomy is crucial for the multimodal treatment of prostate cancer, but limited proof demonstrated enough advantages of the surgery in T4 tumor with bladder invasion. Radical prostatectomy could hardly meet both demands of local tumor control and urinary function. Treatment trends suggest that patients with T4 prostate cancer be treated with radiotherapy combined with androgen deprivation therapy (ADT). However, surgery enables a full pathological assessment of the tumor characteristics and thus a better estimation of the risk of recurrence. Cystoprostatectomy offers an option of surgical treatment for T4 prostate cancer with bladder invasion，which can well remove the bladder and urethra, decrease the risk of positive surgical margins and avoid urination complications.

There is no consensus regarding optimal treatment of T4 prostate cancer and no evidence of oncological outcomes of cystoprostatectomy from clinical trials. A randomized clinical trial comparing two multimodal treatment regimens of cystoprostatectomy and radiotherapy for T4 prostate cancer with bladder invasion is therefore warranted.

DETAILED DESCRIPTION:
1. Determine the subjects

Patients were determined in strict accordance with the inclusion and exclusion criteria, and the trial process and significance were explained to the patients, and informed consent was signed.

2 Randomization

The patients were randomly assigned to surgery group or radiotherapy group according to the random number table.

3 Implementation Process

The intervention measures were divided into operation group and non-operation group. The operation group was given cystoprostatectomy + expanded pelvic lymph node dissection + urinary diversion. The non-operation group received radiotherapy plus androgen deprivation therapy.

4 Follow-up Process

Follow-up was performed once a month (12 times in total) in the first year after surgery or radiotherapy, once every 3 months (4 times in total) in the second year, and once every six months after 2 years. Follow-up items included the presence of complications, digital rectal examination, PSA and testosterone levels, liver and kidney function. If digital rectal examination is positive and serum PSA continues to rise, pelvic MRI and bone scan should be performed. Bone pain, regardless of PSA level, should be scanned.

FunctionalAssessment of Cancer Therapy-General (FACT-G; FunctionalAssessment of Cancer Therapy-Prostate, FACT-P) and color Doppler ultrasonography of bilateral kidney and ureter were performed once every six months after 1 year.

Pelvic MRI, bone scan, chest radiograph, and color ultrasound of abdomen (liver, bile, pancreas and spleen) were examined once a year after surgery or radiotherapy.

Other follow-up examination items or follow-up time can be selected according to special circumstances. The patients were followed up for at least 10 years after surgery or after the end of radiotherapy.

5. Monitoring and management of recurrence, metastasis and complications

If biochemical recurrence after surgery (PSA level two consecutive acuity 0.2 ng/ml, two test interval of 2 weeks) or local recurrence, choose save radiotherapy, 8 Gy single, range is the whole pelvic, continued progress or control again after recurrence after radiotherapy are endocrine therapy, and its solution for than carew amine (50 mg 1 time, 1 times a day, Orally) + Goserelin (3.6mg once every 28 days, subcutaneously injected into the anterior abdominal wall); Patients with extensive metastasis after surgery were treated directly with endocrine therapy (bicalutamide 50mg once daily, orally) plus gosererin (3.6mg once every 28 days, subcutaneously injected into the anterior abdominal wall). The remaining tumor progression was managed according to the recommendations of authoritative guidelines at home and abroad.

The time of occurrence, name of complication, patient status, Clavien-Dindo complication classification, treatment measures and procedures, and treatment results were recorded. Complications were managed according to the recommendations of the guidelines and the experience of our unit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤75, at the time of randomization
2. Newly diagnosed primary prostatic adenocarcinoma confirmed by pathological examination of biopsy；diagnosed within 6 months prior to randomization
3. Untreated for surgery, radiotherapy, or androgen deprivation therapy
4. Eastern Cooperative Oncology Group (ECOG) performance status 0- 2; American Standards Association (ASA) classification I-III
5. A life expectation of at least 10 years
6. Tumor stage (T, M, N): Clinical T4N0M0 with bladder invasion (confirmed by MRI)
7. Eligible for either treatment of cystoprostatectomy or radiotherapy
8. Signed informed consent should be obtained from both the patient or one authorized legal relative.

Exclusion Criteria:

1. Patients with a history of other cancer diagnoses except non-melanoma skin cancer
2. Patients with pelvic surgery
3. Patients with severe systemic diseases
4. severe kidney function -glomerular filtration rate (GFR) < 30 ml/min or elevated liver transaminases above > 10 upper limit of normal (ULN)
5. Patients who are not able comply with scheduled follow-up visits and examinations with the consideration of patients' physical or mental condition

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-06-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 10 years
  The percentage of subjects in a study who have survived at the the endpoint of the observation since randomization or the interval between randomization and death from any cause.

SECONDARY OUTCOMES:
Biochemical progression-free survival (BPFS) | 10 years
  the interval between randomization and biochemical recurrence or death from any cause or the percentage of subjects in a study who have survived without biochemical recurrence at the endpoint of the observation since randomization
Cancer-specific survival (CSS) | 10 years
  the interval between randomization and tumor recurrence, metastasis, or death from any cause, or the percentage of subjects in a study who have survived without tumor recurrence or metastasis at the endpoint of the observation since randomization
Functional Assessment of Cancer Therapy-General (FACT-G) score | 10 years
  This is a score system assessing cancer patients' quality of life, including four aspects of physical status, social status, emotional status and functional status. The total score ranges from 0-108 and a higher score indicates a better outcome.
Functional Assessment of Cancer Therapy-Prostate (FACT-P) score | 10 years
  This is a score system assessing prostate cancer patients' quality of life. The total score ranges from 0-48 and a higher score indicates a better outcome
complications | 10 years
  the complications and the incidence

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Chen, M.D.,Ph.D, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China